CLINICAL TRIAL: NCT05969496
Title: Neoadjuvant Pembrolizumab and Axitinib in Renal Cell Carcinoma With Associated Inferior Vena Cava Tumor Thrombus (NEOPAX)
Brief Title: Neoadjuvant Pembrolizumab and Axitinib in Renal Cell Carcinoma With Inferior Vena Cava Tumor Thrombus
Acronym: NEOPAX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-1669.cc
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Renal Cancer; Kidney Cancer; Renal Cell Carcinoma; Inferior Vena Cava Thrombosis
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Axitinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Pembrolizumab and Axitinib (Experimental): Neoadjuvant therapy with the combination of Pembrolizumab and Axitinib will be given for eligible RCC patients with an IVC TT for a total of 12 weeks. Patients will then undergo imaging with a contrast enhanced, diffusion weighted imaging MRI of the abdomen to evaluate the IVC TT response. A CT chest will also be done to ensure there is no progression of disease. Patients can undergo definitive surgery per treating Urologist within 2 weeks (+/- 7 days) after end of treatment scan.
  Interventions: Drug: Axitinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Axitinib — Axitinib is a potent oral, vascular endothelial growth factor, c-kit and platelet derived growth factor inhibitor.
  Other Names: Inlyta
Drug: Pembrolizumab — Pembrolizumab is a type of immunotherapy. It stimulates the body's immune system to fight cancer cells. Pembrolizumab targets and blocks a protein called PD-1 on the surface of certain immune cells called T-cells. Blocking PD-1 triggers the T-cells to find and kill cancer cells.
  Other Names: Keytruda

SUMMARY:
The primary objective of this study is to evaluate whether the combination of Pembrolizumab and Axitinib given in the neoadjuvant setting can change the Inferior Vena Cava Tumor Thrombus burden. A decrease in the size of the tumor thrombus can potentially lead to decrease in surgical complications, improve patient related health outcomes, and improve long term outcomes such as progression free survival and overall survival.

DETAILED DESCRIPTION:
Patients will receive the combination of Axitinib 5 mg orally twice daily (can be increased to 7 mg twice daily after 2 weeks, and further to 10 mg twice daily as tolerated) and Pembrolizumab 200 mg IV every 21 days. This combination will be given for a total of 12 weeks (4 cycles). A radiographic assessment will be done up to 12 weeks (4 cycles of therapy) to evaluate the primary endpoint of IVC TT response. Patients will undergo a definitive surgery per treating urologist within 2 weeks (+/- 7 days) after the end of treatment scan.

During the course of the trial, patient-related health outcomes using Kidney Cancer validated questionnaires with FKSI-DRS and FKSI-19 will also be obtained. These are validated paper questionnaires that will be given to each patient on study visits while receiving neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision to sign and date the consent form.
* Stated willingness to comply with all study procedures and be available for the duration of the study.
* Participant self-identified gender ages >/= 18 years old is acceptable and appropriate if they meet other inclusion criteria.
* Histologically proven clear cell component RCC.
* An upfront candidate for definitive surgery per treating Urologist.
* Suitable for and willing to undergo nephrectomy (either cytoreductive or with curative intent) per treating urologist.
* T Stage of any of the following: cT3b, cT3c, cT4
* N stage of any of the following: cN0 or cN1
* M stage of any of the following: cM0 or cM1
* ECOG performance status 0 - 2.
* Urinalysis <2+ protein. If dipstick is ≥2+ then a 24-hour urine collection should be performed, and the patient may enter the trial if urinary protein is <2g per 24 hours.
* All participants who have reproductive potential must have a negative serum or urine pregnancy test within a maximum of 14 days prior to starting trial treatment.

Reproductive potential is defined as the following:

* Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy
  * For males with reproductive potential, use effective birth control during treatment with Axitinib and Pembrolizumab is recommended.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to enrollment.
* Has had major surgery within 4 weeks or received radiation therapy within 1 week prior to enrollment to the study.
* Has had prior treatment with any anti-programmed cell death (anti-PD-1) or programmed cell death ligand 1 (PD-L1), or an antibody targeting any other immune-regulatory receptors or mechanisms.
* Has received prior systemic anti-cancer therapy for RCC with vascular endothelial growth factor (VEGF)/VEGF receptors (VEGFR).
* Has a history of severe hypersensitivity reaction (e.g., generalized rash/erythema, hypotension, bronchospasm, angioedema, or anaphylaxis) to Axitinib.
* Has a diagnosis of immunodeficiency OR is receiving a systemic steroid therapy greater than Prednisone 10 mg daily or a steroid equivalent, or any other form of immunosuppressive therapy within 7 days prior to enrollment to the study except in the case of central nervous system (CNS) metastases.
* Has an active autoimmune disease requiring systemic treatment within the past 2 years OR a documented history of clinically severe autoimmune disease. Note: Participants with vitiligo, Sjogren's syndrome, Type 1 diabetes, resolved childhood asthma/atopy, hypothyroidism or adrenal or pituitary insufficiency who are stable on hormone replacement are not excluded.
* Has a known additional malignancy that has progressed or has required active treatment in the last 3 years. Note: Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ such as breast cancer in situ, thyroid cancer (papillary, hurthle cell or follicular), or localized prostate cancer are acceptable if they have undergone potentially curative therapy.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* ALT or AST above 3 times the upper limit of normal
* Has received a live virus vaccine within 30 days of enrollment to the study.
* Active GI bleeding, as evidenced by hematemesis, hematochezia, or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy.
* Intraluminal metastatic lesion with suspected bleeding, inflammatory bowel disease, ulcerative colitis or other GI condition associated with increased risk of perforation.
* Has QT interval corrected for heart rate (QTc) ≥480 msec.
* Has a history of any of the following cardiovascular conditions within 12 months of enrollment to the study:

  * Myocardial infarction
  * Unstable angina pectoris
  * Cardiac angioplasty or stenting
  * Coronary/peripheral artery bypass graft
  * Class III or IV congestive heart failure per New York Heart Association
  * Cerebrovascular accident or transient ischemic attack
* Has poorly controlled hypertension defined as systolic blood pressure (SBP) ≥150 mm Hg and/or diastolic blood pressure (DBP) ≥90 mm Hg on 3 or more dose optimized anti- hypertensive medication.
* Has evidence of inadequate wound healing per treating physician discretion.
* Has active bleeding disorder or other history of significant bleeding episodes within 30 days of enrollment to the study.
* Has current use (within 7 days of enrollment) or anticipated need for treatment with drugs or foods that are known to be strong cytochrome P450 (CYP3A4/5) inhibitors.
* Has current use (within 7 days of enrollment) or anticipated need for treatment with drugs that are known strong CYP3A4/5 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort; or drugs that are known with proarrhythmic potential.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study by subject self-report.
* Has had a prior solid organ transplant.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate Change in IVC Tumor Thrombus Extent Based on the Mayo Classification | baseline and 12 weeks
  * Patients will get baseline imaging with an MRI of the abdomen to evaluate the level of the IVC TT based on the Mayo Classification. Patients will get an end of treatment MRI at 12 weeks to evaluate the efficacy of neoadjuvant therapy with Pembrolizumab and Axitinib. The Mayo classification is described as below:
  * Level 0: thrombus limited to the renal vein
  * Level 1: into IVC <2cm from renal vein ostium level
  * Level 2: IVC extension >2cm from renal vein ostium and below hepatic vein
  * Level 3: thrombus at the level of or above the hepatic veins but below the diaphragm
  * Level 4: thrombus extending above the diaphragm
Evaluate a change in IVC TT Size from Baseline | baseline and 12 weeks
  o Evaluation of IVC TT anteroposterior and transverse diameter will also be measured at baseline and the end of treatment at 12 weeks. The baseline largest diameter will be subtracted to the largest diameter as the end of treatment divided by the baseline largest diameter will be computed to evaluate the percentage change in the IVC TT size.

SECONDARY OUTCOMES:
Evaluate Surgical Complications after the Neoadjuvant Combination of Pembrolizumab and Axitinib Among Patients with RCC with IVC TT | Date of surgery up to 30 days post operative or date of hospital discharge whichever occurs first
  * Surgical morbidity will be graded based on the Clavien- Dindo Classification. This will be graded as below:
  * Grade I: Any deviation from the normal post-operative course not requiring surgical, endoscopic, or radiological intervention (inc. certain drugs, physiotherapy and wound infections that are opened at the bedside)
  * Grade II: Complications requiring drug treatments other than those allowed for Grade I complications (inc. blood transfusion and total parenteral nutrition (TPN))
  * Grade III: Complications requiring surgical, endoscopic, or radiological intervention (IIIa=not under general anesthetic/IIIb=under general anesthetic)
  * Grade IV: Life-threatening complications (inc. CNS complications requiring intensive care, but excludes transient ischemic attacks (TIAs)) (IVa=single-organ dysfunction (inc. dialysis)/IVb=multi-organ dysfunction)
  * Grade V: Death of the patient
Safety profile of the combination of Axitinib and Pembrolizumab | baseline to 30 days post operative
  Catalogue o Any grade adverse event
  o Grade 3 or higher adverse event possibly, probably, or definitely related to study therapy All treatment related adverse events will be assessed using the Common Terminology Criteria for Adverse Events v5.0
1 year Progression Free Survival | baseline, 3 months, 6 months, 9 months, 12 months from study enrollment
  Progression-free survival is defined as any clinical or radiographic progression or death from any cause one year after enrollment in the study
1 year Overall Survival | 12 months from study enrollment
  One year- Overall survival. Overall survival is defined as death from any cause one year after enrollment in the study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Kessler, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Hilands Ranch Hospital, Highlands Ranch, Colorado
  - Lone Tree Medical Center, Lone Tree, Colorado

IPD SHARING:
Plan to Share IPD: No